CLINICAL TRIAL: NCT04228874
Title: The Short Term Effect of Stent Size and Number on Left Ventricular Mechanical Dyssynchrony After Elective PCI to Left Anterior Descending Artery
Brief Title: Effect of Stent Size on Dyssynchrony
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, shaimaa Mostafa, assistant professor, Benha University
Other Study IDs: dyssynchrony
Record Dates: First submitted 2019-12-19; First posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Left Ventricular Function
Keywords: Stent length; Stent diameter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: coronary artery stents — Coronary angiography was done for all the patients according to the Judkins technique. All images were evaluated by an experienced operator, significant coronary artery disease was defined as > 70 % luminar diameter stenos. The following data was obtained:
  * Site of stent implantation within LAD. The first Diagonal branch serves as the boundary between the proximal and mid portion of the LAD. Thus, the portion of the artery prior to the origin of the 1st diagonal is known as the proximal LAD, while the segment just below the1st diagonal branch is the mid LAD. The distal segment of the LAD is the terminal third of the artery (Cao et al., 2017).
  * Length, diameter and number of stents.
  * TIMI flow after stent deployment.

SUMMARY:
the effect of stent size and number on left ventricular mechanical dyssynchrony after PCI using drug eluting stent is not clear enough

DETAILED DESCRIPTION:
Background: the effect of stent size and number on left ventricular mechanical dyssynchrony after PCI using drug eluting stent is not clear enough Aim: to study short term effect of stent size and number on left ventricular mechanical dyssynchrony after elective PCI to LAD artery.

Patients and methods: the study included 150 adult patients with electively stented LAD lesion with DES. Patients were evaluated pre PCI then follow up at 1m and 3m using tissue synchronization image (TSI).

ELIGIBILITY:
Inclusion Criteria:

* adult patients with electively stented LAD lesion with DES were enrolled in the study. Patients were evaluated pre PCI then follow up at 1m and 3m after PCI using TSI.

Exclusion Criteria:

* patients with Bundle branch block (BBB),
* Previous percutaneous coronary intervention (PCI),
* Previous coronary artery bypass graft (CABG),
* Rhythm other than sinus,
* Rheumatic heart disease,
* Prosthetic valve,
* Complicated or unsuccessful procedure,
* Patients with significant degenerative changes,
* Patients with previous STEMI,
* and dropped patients from follow up were excluded from the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with electively stented LAD lesion with DES were enrolled in the study
Sampling Method: Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
left ventricular systolic function | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- shaimaa Mostafa, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
included in the research